CLINICAL TRIAL: NCT01955824
Title: "A RCT ON CLINICAL EFFICACY OF 1% vs. 2% LIGNOCAINE IN COUGH SUPPRESSION AND PAIN RELIEF IN PATIENTS UNDERGOING FLEXIBLE BRONCHOSCOPY"
Brief Title: A Trial on Clinical Efficacy of 1% Versus 2% Lignocaine in Cough Suppression and Pain Relief in Patients Undergoing Flexible Bronchoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bron/Lig/Tr-1
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Lung Cancer; Tuberculosis; Sarcoidosis; Interstitial Lung Disease
Keywords: bronchoscopy; lignocaine; cough
MeSH Terms: conditions — Lung Neoplasms; Tuberculosis; Sarcoidosis; Lung Diseases, Interstitial; Cough | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1% lignocaine (Experimental): Each patient included in study will be nebulized prior to flexible bronchoscopy with 2.5 ml of 4% lignocaine. This will be followed by spray of 2 puffs of 10% lignocaine over the posterior pharynx and vocal cords. Lignocaine jelly (2%) will be applied in the nasal cavity. Lignocaine (1%) 8ml will be administered as "spray as you go" technique through the bronchoscope over the vocal cords, carina, right and left main bronchus as aliquots of 2 ml each. Additional requirement of lignocaine will also be recorded for all the patients.
  Interventions: Drug: 1% lignocaine
- 2% lignocaine (Active Comparator): Each patient included in study will be nebulized prior to flexible bronchoscopy with 2.5 ml of 4% lignocaine. This will be followed by spray of 2 puffs of 10% lignocaine over the posterior pharynx and vocal cords. Lignocaine jelly (2%) will be applied in the nasal cavity. Lignocaine (2%) 8ml will be administered as "spray as you go" technique through the bronchoscope over the vocal cords, carina, right and left main bronchus as aliquots of 2 ml each. Additional requirement of lignocaine will also be recorded for all the patients.
  Interventions: Drug: 2% lignocaine

INTERVENTIONS:
Drug: 1% lignocaine
  Arms: 1% lignocaine
Drug: 2% lignocaine
  Arms: 2% lignocaine

SUMMARY:
Flexible bronchoscopy is a common procedure performed by pulmonary physicians. The use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy varies among physicians, institutions and geographic locations across the globe. Commonly used topical anesthetic agents before and during bronchoscopy include cocaine (4%),benzocaine (20%), tetracaine (1%), and lignocaine (1%-10%). Topical lignocaine is administered through the flexible bronchoscope in an attempt to reduce excessive coughing and patient discomfort. However, the optimal dosage and strength of topical lignocaine that should be used during fibreoptic bronchoscopy has long been a topic of controversy. In this study we compare the efficacy of 1% versus 2% lignocaine in controlling cough and pain in patients undergoing flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing flexible bronchoscopy
* Hemodynamic stability

Exclusion Criteria:

* Patients receiving sedatives during the course of their treatment
* Patients undergoing conventional TBNA and/or EBUS-TBNA who are likely to receive sedation
* Patients with known hypersensitivity to lignocaine
* Not willing to provide informed consent

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cough suppression (by Operator and Patient) | 15 minutes
  Cough will be rated on a visual analog scale (VAS) from 0 (no cough) to 100 mm (worst cough ever)
Pain control | 15 minutes
  Pain will be assessed on Wong Baker Face rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Bronchoscopy suite, PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Kaur H, Dhooria S, Aggarwal AN, Gupta D, Behera D, Agarwal R. A Randomized Trial of 1% vs 2% Lignocaine by the Spray-as-You-Go Technique for Topical Anesthesia During Flexible Bronchoscopy. Chest. 2015 Sep;148(3):739-745. doi: 10.1378/chest.15-0022. PMID 25811287